CLINICAL TRIAL: NCT01953640
Title: PROstate Cancer Medically Optimized Genome Enhanced ThErapy (PROMOTE)
Brief Title: Gene Expression in Patients With Metastatic Prostate Cancer Receiving CYP-17 Inhibition Therapy
Acronym: PROMOTE
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: MC1351; R01CA130908 (NIH); R01CA212097 (NIH); R01CA203849 (NIH); W81XWH-15-1-0634 (Other Grant/Funding Number: Department of Defense); NCI-2013-01628 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13-001296 (Other: Mayo Clinic Institutional Review Board); MC1351 (Other: Mayo Clinic)
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Hormone-Resistant Prostate Cancer; Metastatic Prostate Carcinoma; Prostate Adenocarcinoma; Recurrent Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with DNA and RNA will be retained.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-correlative (gene expression with CYP-17 inhibition): Laboratory Biomarker Analysis: Tissue, blood, and urine samples are collected at baseline and after 12-14 weeks of treatment and assessed for circulating tumor cells, genome-wide SNP, and exome sequencing. Subjects will also receive a Quality-of-Life Assessment.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This research trial studies gene expression in patients with prostate cancer that has spread to other places in the body receiving cytochrome P450 17 alpha hydroxylase/17,20 lyase (CYP-17) inhibition therapy. Studying samples of tissue, blood, and urine in the laboratory from patients receiving CYP-17 inhibition therapy may help doctors learn more about changes that occur in deoxyribonucleic acid (DNA) and identify biomarkers related to cancer. It may also help doctors understand how well patients respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether somatic tumor genome alterations identified in tumor tissue before or after the initiation of CYP-17 inhibition with abiraterone acetate therapy are associated with a 12-week composite progression free survival (PFS) endpoint.

II. To use tumor tissue obtained prior to the initiation of therapy and from the 12 week biopsy to develop tumor xenografts for mechanistic and functional studies which will determine whether mutations identified in the tumor genome are associated with response to drugs that target the observed mutated genes and/or associated pathways.

SECONDARY OBJECTIVES:

I. To determine whether somatic tumor genome alterations identified before or after initiating CYP-17 inhibition with abiraterone acetate therapy are associated with overall survival.

II. To determine whether somatic tumor genome alterations identified in tumor tissue before or after the initiation of CYP-17 inhibition with abiraterone acetate therapy are associated with progression free survival (PFS).

III. To evaluate circulatory markers in blood and urine specimens for response and/or resistance to treatment. (Exploratory and correlative objectives)

OUTLINE:

Tissue, blood, and urine samples are collected at baseline and after 12-14 weeks of treatment and assessed for circulating tumor cells, genome-wide single-nucleotide polymorphism (SNP), and exome sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of adenocarcinoma of the prostate or documented history in medical records of having received treatment for prostate cancer diagnosis
* Metastatic disease on chest, abdominal, or pelvic computed tomography (CT) and/or bone scan amenable to biopsy
* Hemoglobin (HgB) > 9.0 gm
* Absolute neutrophil count (ANC) >= 1500 cells/L
* Platelets >= 100,000 u/L
* Creatinine =< 1.5 x upper limit of normal (ULN)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase (AST)) and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase (ALT)) =< 1.5 x ULN
* Castrate serum testosterone level (< 50 ng/dL -or- < 1.7 nmol/L)
* Progression while on or after androgen deprivation therapy defined as:

  * Progressive measurable disease: at least a 20% increase in the sum of the longest diameters of measurable lesions over the smallest sum observed or the appearance of one or more new lesions as assessed by imaging during hormone ablation treatment; measurable lesions are nodal or visceral soft-tissue lesions with nodal lesions >= 20 mm in diameter or visceral/soft-tissue lesions >= 10 mm in diameter OR
  * Bone scan progression: appearance of 2 or more new lesions on bone scan during hormone ablation treatment OR
  * Increasing serum prostate-specific antigen (PSA) level: two consecutive increases in PSA levels documented over a previous reference value obtained at least one week apart are required; if the third PSA value is less than the second, an additional fourth test to confirm a rising PSA is acceptable; a minimum starting value of 2.0 ng/mL is required for study enrollment
  * Note: androgen deprivation therapy may have included either medical or surgical castration
* >= 14 days has passed since completing radiotherapy (exception for radiotherapy: >= 7 days since completing a single fraction of =< 800 centigray (cGy) to a restricted field or limited-field radiotherapy to non-marrow bearing area such as an extremity or orbit) at the time of registration
* Patients who may have received systemic chemotherapy or any novel therapeutic CYP-17 inhibitor and/or novel androgen receptor (AR) inhibitor agents previously for prostate cancer should have received the last dose of the previously administered systemic therapy >= 12 months from the date of registration
* Provide informed written consent
* Has recovered from any other therapy-related toxicity to =< grade 2, (except alopecia, anemia and any signs or symptoms of androgen deprivation therapy)
* Willing to provide tissue and blood samples for correlative research purposes
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Patient is considered a candidate for initiating CYP-17 inhibitors abiraterone acetate and prednisone after failure of hormonal therapy and has no contra-indication to starting this combination as standard of care
* Patients have stopped any antiandrogen therapy (including bicalutamide) >= 4 weeks prior to first dose of study drug; in addition any other therapies for prostate cancer, other than gonadotropin-releasing hormone (GnRH) analogue therapy, such as progesterone, medroxyprogesterone, progestins (megestrol), or 5-alpha reductase inhibitors (e.g., finasteride or dutasteride), must be discontinued >= 2 weeks before the first dose of study drug

Exclusion Criteria:

* Use of any of these therapies =< 12 months prior to registration:

  * Use of any of the standard therapies for castrate resistant prostate cancer (CRPC) stage =< 12 months prior to registration; Note: see below for further exclusion details of specific standard therapies

    * Initiation of full dose chemotherapy with docetaxel for CRPC stage =< 12 months prior to registration is an exclusion criterion

      * Note: docetaxel for hormone sensitive prostate cancer is not an exclusion criterion
    * Use of radium-223 for CRPC stage is an exclusion criteria
    * Use of Provenge vaccine for CRPC =< 12 months prior to registration is an exclusion criterion

      * Note: less than 3 doses of Provenge vaccine =< 12 months prior to registration for CRPC is not an exclusion criterion
    * Initiation of full dose chemotherapy with mitoxantrone for CRPC stage with-in the previous 12 months is an exclusion criterion
    * Use of cabazitaxel chemotherapy =< 12 months prior to registration is an exclusion criterion

      * Note: initiation of full dose chemotherapy with cabazitaxel for CRPC stage with-in the previous 12 months is an exclusion criterion
    * Use of ketoconazole with steroids =< 12 months prior to registration for CRPC stage

      * Note: ketoconazole therapy taken for a time period of =< 12 weeks in the 12 month period prior to registration is not an exclusion criterion
    * Use of enzalutamide for CRPC stage =< 12 months prior to registration is an exclusion criteria use of any experimental or standard of care CYP-17 inhibitors =< 12 months prior to registration is an exclusion criteria

      * Note: standard of care CRPC therapy with a CYP-17 inhibitor =< 7 days prior to registration is not an exclusion criterion; if taken for 8 days or more it will be counted as an exclusion criterion
* Receiving any intermittent hormonal treatment GnRH analogues and has not yet achieved sub-castrate levels of testosterone (< 50 ng/dl or < 1.7 mmol/L)
* History of or current documented brain metastasis or carcinomatous meningitis, treated or untreated; Note: brain imaging for asymptomatic patients is not required
* Current symptomatic cord compression requiring surgery or radiation therapy

  * Note: once successfully treated and there has been no progression, patients are eligible for the study
* Active second malignancy (except non-melanomatous skin or superficial bladder cancer) defined as requiring anticancer therapy or at high risk of recurrence during the study
* Uncontrolled medical conditions such as heart failure, myocardial infarction, uncontrolled hypertension, disseminated on-going coagulopathy, stroke or treatment of a major active infection =< 3 months of registration, as well as any significant concurrent medical illness that in the opinion of the Investigator would preclude protocol therapy
* Planned concomitant participation in another clinical trial of an experimental agent, vaccine, or device

  * Note: concomitant participation in observational studies is acceptable
* Patients with a global or severe deterioration of health status such that it requires discontinuation of standard of care treatments for CRPC stage without evidence of disease progression =< 12 weeks prior to registration

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males age > 18 years with adenocarcinoma of the prostate
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2013-05-30 (Actual); Primary Completion 2015-12-03 (Actual); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Occurrence of PFS as defined by Prostate Cancer Working Group 2 criteria | Up to 14 weeks

SECONDARY OUTCOMES:
Overall survival after receiving abiraterone acetate | Up to 5 years
  Kaplan-Meier curve and Cox proportional hazard regression model will be used to summarize overall survival until 5 years after abiraterone therapy in this trial.
PFS after receiving abiraterone acetate | Up to 5 years

OTHER OUTCOMES:
Circulating tumor cells | Up to 14 weeks
  Descriptive statistics and graphical procedures will be used for summarizing circulating tumor cells. The quantity of circulating tumor cells at baseline and after abiraterone therapy will be correlated with PFS at 12-14 weeks.
Novel somatic changes within gene and gene pathway that form the genomic signature | Baseline to up to 14 weeks
Tumor "signatures" by using immortalized xenograft models | Up to 14 weeks
  Descriptive statistics and graphical procedures will be used for summarizing "tumor signature" for xenograft model. The results of xenograft model will be correlated with PFS at 12-14 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Winston Tan, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qin S, Liu D, Kohli M, Wang L, Vedell PT, Hillman DW, Niu N, Yu J, Weinshilboum RM, Wang L. TSPYL Family Regulates CYP17A1 and CYP3A4 Expression: Potential Mechanism Contributing to Abiraterone Response in Metastatic Castration-Resistant Prostate Cancer. Clin Pharmacol Ther. 2018 Jul;104(1):201-210. doi: 10.1002/cpt.907. Epub 2017 Nov 22. PMID 29027195
- [Derived] Hart SN, Ellingson MS, Schahl K, Vedell PT, Carlson RE, Sinnwell JP, Barman P, Sicotte H, Eckel-Passow JE, Wang L, Kalari KR, Qin R, Kruisselbrink TM, Jimenez RE, Bryce AH, Tan W, Weinshilboum R, Wang L, Kohli M. Determining the frequency of pathogenic germline variants from exome sequencing in patients with castrate-resistant prostate cancer. BMJ Open. 2016 Apr 15;6(4):e010332. doi: 10.1136/bmjopen-2015-010332. PMID 27084275
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials